CLINICAL TRIAL: NCT02227862
Title: An Open-Label, Randomized, Multi-Center, Parallel-Group Clinical Trial Comparing the Efficacy and Safety of Mylan's Insulin Glargine With Lantus® in Type 1 Diabetes Mellitus Patients
Brief Title: Non-inferiority Study to Compare the Efficacy and Safety of Mylan's Insulin Glargine With Lantus® in Type 1 Diabetes Mellitus Patients (INSTRIDE 1)
Acronym: INSTRIDE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Mylan GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYL-GAI-3001
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Results first posted 2020-03-09 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mylan's Insulin Glargine (Experimental): Receive Mylan's Insulin Glargine plus insulin lispro.
  Interventions: Drug: Mylan's insulin glargine
- Lantus® (Active Comparator): Receive Lantus® plus insulin lispro
  Interventions: Drug: Lantus®

INTERVENTIONS:
Drug: Mylan's insulin glargine — All patients will be shifted from their current mealtime insulin to insulin lispro at the start of the run-in period, and will continue on this for the complete trial. During the 6 week run-in period the doses of Lantus® and insulin lispro will be titrated (if required) to ensure diabetes control. After the run-in period, patients will be randomized to receive either Mylan's insulin glargine (in place of Lantus®), or to continue on Lantus®. During the period from 12 to 24 weeks dose titration will be kept to a minimum.
  Arms: Mylan's Insulin Glargine
Drug: Lantus® — All patients will be shifted from their current mealtime insulin to insulin lispro at the start of the run-in period; and will continue on this for the complete trial. During the 6week run-in period the doses of Lantus® and insulin lispro will be titrated (if required) to ensure diabetes control. After the run-in period, patients will be randomized to receive either Mylan's insulin glargine (in place of Lantus®), or to continue on Lantus®. During the period from 12 to 24 weeks dose titration will be kept to a minimum.
  Arms: Lantus®

SUMMARY:
To test whether Mylan's insulin glargine once daily is non-inferior to Lantus® once daily (based on change in HbA1c from baseline to 24 weeks) when administered in combination with mealtime insulin lispro.

DETAILED DESCRIPTION:
This trial is a multicenter, open-label, randomized, parallel-group trial in patients with Type 1 Diabetes Mellitus (T1DM) comparing the efficacy and safety of Mylan's insulin glargine with that of Lantus®.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an established diagnosis of T1DM per ADA 2014 criteria
* Body mass index (BMI) of 18.5 to 35 kg/m2 at screening (both values inclusive).
* Glycosylated hemoglobin (HbA1c) ≤9.5% at screening.
* Hemoglobin ≥9.0 g/dL at screening.

Exclusion Criteria:

* History of hypersensitivity to any of the active or inactive ingredients of the insulin/insulin analogue preparations used in the trial, OR history of significant allergic drug reactions.
* History of use of animal insulin within the last 3 years or use of biosimilar insulin glargine at any time prior.
* History of use of a regular immunomodulator therapy in the 1 year prior to screening.
* History of ≥2 episodes of severe hypoglycemia within the 6 months before screening or history of hypoglycemia unawareness (a sample questionnaire is provided in Appendix I), as judged by the investigator.
* History of ≥1 episodes of diabetic ketoacidosis or emergency room visits for uncontrolled diabetes leading to hospitalization within the 6 months prior to screening.
* Serological evidence of human immunodeficiency virus (HIV), hepatitis B (HbSAg) or hepatitis C (HCVAb) antibodies at screening.
* History of drug or alcohol dependence or abuse during the 1 year prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Blevins, MD, Principal Investigator — Texas Diabetes & Endocrinology
Locations (143):
- United States (68):
  - Mylan Investigational Site, Bell Gardens, California
  - Mylan Investigational Site, Fresno, California
  - Mylan Investigational Site, Greenbrae, California
  - Mylan Investigational Site, La Jolla, California
  - Mylan Investigational Site, La Mesa, California
  - Mylan Investigational Site, Long Beach, California
  - Mylan Investigational Site, Los Gatos, California
  - Mylan Investigational Site, Mission Hills, California
  - Mylan Investigational Site, National City, California
  - Mylan Investigational Site, Northridge, California
  - Mylan Investigational Site, Tustin, California
  - Mylan Investigational Site, Walnut Creek, California
  - Mylan Investigational Site, Bradenton, Florida
  - Mylan Investigational Site, Cooper City, Florida
  - Mylan Investigational Site, Hialeah, Florida
  - Mylan Investigational Site, Hollywood, Florida
  - Mylan Investigational Site, Miami, Florida
  - Mylan Investigational Site, New Port Richey, Florida
  - Mylan Investigational Site, Palm Harbor, Florida
  - Mylan Investigational Site, West Palm Beach, Florida
  - Mylan Investigational Site, Atlanta, Georgia
  - Mylan Investigational Site, Columbus, Georgia
  - Mylan Investigational Site, Honolulu, Hawaii
  - Mylan Investigational Site, Idaho Falls, Idaho
  - Mylan Investigational Site, Crystal Lake, Illinois
  - Mylan Investigational Site, LaGrange, Illinois
  - Mylan Investigational Site, Springfield, Illinois
  - Mylan Investigational Site, Anderson, Indiana
  - Mylan Investigational Site, Muncie, Indiana
  - Mylan Investigational Site, Council Bluffs, Iowa
  - Mylan Investigational Site, Des Moines, Iowa
  - Mylan Investigational Site, Overland Park, Kansas
  - Mylan Investigational Site, Topeka, Kansas
  - Mylan Investigational Site, Lexington, Kentucky
  - Mylan Investigational Site, Billings, Montana
  - Mylan Investigational Site, Omaha, Nebraska
  - Mylan Investigational Site, Las Vegas, Nevada
  - Mylan Investigational Site, Albany, New York
  - Mylan Investigational Site, Mineola, New York
  - Mylan Investigational Site, Staten Island, New York
  - Mylan Investigational Site, Syracuse, New York
  - Mylan Investigational Site, Asheville, North Carolina
  - Mylan Investigational Site, Burlington, North Carolina
  - Mylan Investigational Site, Greensboro, North Carolina
  - Mylan Investigational Site, Greenville, North Carolina
  - Mylan Investigational Site, Hickory, North Carolina
  - Mylan Investigational Site, Morehead City, North Carolina
  - Mylan Investigational Site, Wilmington, North Carolina
  - Mylan Investigational Site, Cincinnati, Ohio
  - Mylan Investigational Site, Mentor, Ohio
  - Mylan Investigational Site, Bend, Oregon
  - Mylan Investigational Site, Corvallis, Oregon
  - Mylan Investigational Site, Chattanooga, Tennessee
  - Mylan Investigational Site, Memphis, Tennessee
  - Mylan Investigational Site, Austin, Texas
  - Mylan Investigational Site, Dallas, Texas
  - Mylan Investigational Site, El Paso, Texas
  - Mylan Investigational Site, Round Rock, Texas
  - Texas Diabetes & Endocrinology, Round Rock, Texas
  - Mylan Investigational Site, San Antonio, Texas
  - Mylan Investigational Site, Ogden, Utah
  - Mylan Investigational Site, Salt Lake City, Utah
  - Mylan Investigational Site, South Jordan, Utah
  - Mylan Investigational Site, Chesapeake, Virginia
  - Mylan Investigational Site, Manassas, Virginia
  - Mylan Investigational Site, Renton, Washington
  - Mylan Investigational Site, Tacoma, Washington
  - Mylan Investigational Site, Vancouver, Washington
- Canada (6):
  - Mylan Investigational Site, Red Deer, Alberta
  - Mylan Investigational Site, Vancouver, British Columbia
  - Mylan Investigational Site, Winnipeg, Manitoba
  - Mylan Investigational Site, Laval, Quebec
  - Mylan Investigational Site, Mirabel, Quebec
  - Mylan Investigational Site, Montreal, Quebec
- Czechia (7):
  - Mylan Investigational Site, Brno
  - Mylan Investigational Site, Broumov
  - Mylan Investigational Site, Bruntál
  - Mylan Investigational Site, České Budějovice
  - Mylan Investigational Site, Olomouc
  - Mylan Investigational Site, Pardubice
  - Mylan Investigational Site, Prague
- Estonia (3):
  - Mylan Investigational Site, Pärnu
  - Mylan Investigational Site, Tallinn
  - Mylan Investigational Site, Tartu
- Germany (9):
  - Mylan Investigational Site, Hohenmölsen, Anhalt
  - Mylan Investigational Site, Wangen, Baden-Wurttemberg
  - Mylan Investigational Site, Aschaffenburg, Bavaria
  - Mylan Investigational Site, Schweinfurt, Bavaria
  - Mylan Investigational Site, Frankfurt am Main, Hesse
  - Mylan Investigational Site, Münster, North Rhine-Westphalia
  - Mylan Investigational Site, Sankt Ingbert, Saarland
  - Mylan Investigational Site, Dresden, Saxony
  - Mylan Investigational Site, Hamburg
- Hungary (8):
  - Mylan Investigational Site, Baja
  - Mylan Investigational Site, Budapest
  - Mylan Investigational Site, Eger
  - Mylan Investigational Site, Gyula
  - Mylan Investigational Site, Létavértes
  - Mylan Investigational Site, Makó
  - Mylan Investigational Site, Miskolc
  - Mylan Investigational Site, Szeged
- Latvia (6):
  - Mylan Investigational Site, Kuldīga
  - Mylan Investigational Site, Limbaži
  - Mylan Investigational Site, Ogre
  - Mylan Investigational Site, Riga
  - Mylan Investigational Site, Sigulda
  - Mylan Investigational Site, Talsi
- Romania (9):
  - Mylan Investigational Site, Bacau
  - Mylan Investigational Site, Baia Mare
  - Mylan Investigational Site, Bucharest
  - Mylan Investigational Site, Buzău
  - Mylan Investigational Site, Cluj-Napoca
  - Mylan Investigational Site, Galati
  - Mylan Investigational Site, Iași
  - Mylan Investigational Site, Oradea
  - Mylan Investigational Site, Timișoara
- Slovakia (18):
  - Mylan Investigational Site, Banská Bystrica
  - Mylan Investigational Site, Bardejov
  - Mylan Investigational Site, Bratislava
  - Mylan Investigational Site, Dolný Kubín
  - Mylan Investigational Site, Košice
  - Mylan Investigational Site, Levice
  - Mylan Investigational Site, Ľubochňa
  - Mylan Investigational Site, Nové Mesto nad Váhom
  - Mylan Investigational Site, Nové Zámky
  - Mylan Investigational Site, Prešov
  - Mylan Investigational Site, Prievidza
  - Mylan Investigational Site, Pruské
  - Mylan Investigational Site, Rimavská Sobota
  - Mylan Investigational Site, Sabinov
  - Mylan Investigational Site, Skalica
  - Mylan Investigational Site, Štúrovo
  - Mylan Investigational Site, Trebišov
  - Mylan Investigational Site, Žilina
- South Africa (6):
  - Mylan Investigational Site, Bloemfontein, Free State
  - Mylan Investigational Site, Johannesburg, Gauteng
  - Mylan Investigational Site, Krugersdorp, Gauteng
  - Mylan Investigational Site, Pretoria, Gauteng
  - Mylan Investigational Site, Durban, KwaZulu-Natal
  - Mylan Investigational Site, Cape Town, Western Cape
- United Kingdom (3):
  - Mylan Investigational Site, Plymouth, Devon
  - Mylan Investigational Site, Leicester, Leicestershire
  - Mylan Investigational Site, Swansea

REFERENCES:
- [Derived] Sun B, Sengupta N, Rao A, Donnelly C, Waichale V, Roy AS, Ramaswamy S, Pathak D, Bowsher RR, Raiter Y, Aubonnet P, Barve A. Similar immunogenicity profiles between the proposed biosimilar MYL-1501D and reference insulin glargine in patients with diabetes mellitus: the phase 3 INSTRIDE 1 and INSTRIDE 2 studies. BMC Endocr Disord. 2021 Jun 26;21(1):129. doi: 10.1186/s12902-021-00797-4. PMID 34174848

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mylan's Insulin Glargine | Lantus®
Started | 280 | 278
Week 24 | 269 | 263
Completed | 261 | 256
Not Completed | 19 | 22
Not completed — Protocol Violation | 7 | 9
Not completed — Other | 0 | 2
Not completed — Adverse Event | 4 | 3
Not completed — Withdrawal by Subject | 7 | 6
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mylan's Insulin Glargine | Lantus® | Total
Number analyzed (Participants) | 280 | 278 | 558
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 275 | 272 | 547
  >=65 years | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12.03) | 42.2 (11.97) | 42.1 (11.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 106 | 222
  Male | 164 | 172 | 336
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 2 | 4
  Black | 2 | 5 | 7
  Caucasian | 263 | 265 | 528
  Hispanic | 6 | 3 | 9
  Other | 7 | 3 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  Europe | 145 | 145 | 290
  North America | 126 | 126 | 252
  South Africa | 9 | 7 | 16
Insulin History [Count of Participants; unit: Participants]
  Yes | 280 | 277 | 557
  No | 0 | 1 | 1
Dosing Time [Count of Participants; unit: Participants]
  Morning | 38 | 40 | 78
  Evening | 242 | 238 | 480
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 26.435 (3.7058) | 26.636 (4.2022) | 26.535 (3.9586)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 18.685 (11.7771) | 19.697 (11.2868) | 19.206 (11.5411)
Baseline fasting plasma glucose [Mean (Standard Deviation); unit: mg/dL] | 167.4 (68.43) | 163.9 (61.61) | 165.6 (65.09)
Baseline HbA1c [Mean (Standard Deviation); unit: percent] | 7.37 (0.869) | 7.39 (0.843) | 7.38 (0.855)
Baseline fasting C-peptide [Mean (Standard Deviation); unit: mmol/L] | 0.298 (0.2291) | 0.291 (0.2508) | 0.295 (0.2395)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to 24 Weeks
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 280 | 277
percent | 0.14 (0.054) | 0.11 (0.054)

2. Secondary Outcome: Summary of Actual and Change From Baseline in HbA1c
Time Frame: 24 and 52 weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 280 | 277
percent
  week 24 | 0.12 (0.599) | 0.09 (0.526)
  week 52 | 0.2 (0.633) | 0.25 (0.595)

3. Secondary Outcome: Change From Baseline in FPG Over Time
Time Frame: 24 and 52 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 280 | 277
mmol/L
  week 24 | -0.81 (4.485) | 0.09 (4.507)
  week 52 | 0.23 (4.281) | 0.43 (4.455)

4. Secondary Outcome: Change From Baseline in 8-point SMBG Profile Over Time
Time Frame: 24 and 52 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 280 | 277
mmol/L
  week 24 | 0.038 (2.3751) | -0.095 (1.5012)
  week 52 | -0.082 (1.5032) | -0.082 (1.5267)

5. Secondary Outcome: Change in Total Daily Insulin Dose Per Unit Body Weight From Baseline Over Time
Time Frame: 24 and 52 weeks
Measure: Mean (Standard Deviation); unit: U/Kg
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 280 | 277
U/Kg
  week 24 | 0.0203 (0.09962) | 0.0127 (0.10871)
  week 52 | 0.0278 (0.1044) | 0.0138 (0.11372)

6. Secondary Outcome: Rate of Hypoglycemic Events Per 30 Days Over Time
Time Frame: 24 and 52 weeks
Measure: Mean (Standard Deviation); unit: Episodes/30 Days
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 280 | 278
Episodes/30 Days
  week 24 | -5.162 (9.0724) | -4.93 (8.3815)
  week 52 | -6.241 (9.214) | -5.765 (8.3658)

7. Secondary Outcome: Hypoglycemia Occurrence
Time Frame: 52 weeks
Measure: Number; unit: Number of patients
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 280 | 278
Number of patients
  Any hypoglycemic event | 273 | 269
  Severe hypoglycemia | 11 | 13
  Documented symptomatic hypoglycemia | 249 | 249
  Asymptomatic hypoglycemia | 246 | 243
  Probable symptomatic hypoglycemia | 37 | 36
  Relative hypoglycemia | 35 | 44
  Other hypoglycemia | 19 | 19
  Unknown | 77 | 71

8. Secondary Outcome: Occurrence of Local and Systematic Reactions
Time Frame: 52 weeks
Measure: Number; unit: Number of patients
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 280 | 278
Number of patients
  Local | 3 | 4
  Systemic | 2 | 2

9. Secondary Outcome: Change in Total Insulin Antibody Percent Binding for Mylan's Insulin Glargine Assay Over Time
Time Frame: 24 and 52 weeks
Measure: Mean (Standard Deviation); unit: %SB
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 280 | 278
%SB
  week 24 | -0.3063 (7.22075) | 0.3592 (7.16624)
  week 52 | -0.9591 (8.51754) | -1.0634 (8.42794)

10. Secondary Outcome: Change in Total Insulin Antibody Percent Binding for Lantus Assay Over Time
Time Frame: 24 and 52 weeks
Measure: Mean (Standard Deviation); unit: %SB
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 280 | 278
%SB
  week 24 | -0.215 (7.3298) | 0.157 (7.411)
  week 52 | -0.896 (8.5610) | -1.233 (8.623)

11. Secondary Outcome: Change in Cross-reactive Insulin Antibody Percent Binding for Mylan's Insulin Glargine Assay Over Time
Time Frame: 24 and 52 weeks
Measure: Mean (Standard Deviation); unit: %SB
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 280 | 278
%SB
  week 24 | -0.363 (7.1081) | 0.27 (7.1204)
  week 52 | -1.132 (8.3911) | -1.21 (8.4096)

12. Secondary Outcome: Change in Cross-reactive Insulin Antibody Percent Binding for Lantus Assay Over Time
Time Frame: 24 and 52 weeks
Measure: Mean (Standard Deviation); unit: %SB
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 280 | 278
%SB
  week 24 | -0.265 (7.2543) | 0.055 (7.3985)
  week 52 | -1.060 (8.4414) | -1.367 (8.6848)

13. Secondary Outcome: Proportion of Patients With HbA1c < 7%
Time Frame: 24 and 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 280 | 277
Participants
  week 24 | 73 | 84
  week 52 | 65 | 61

ADVERSE EVENTS:
Time Frame: 56 Weeks
Description: After Week 52, all the patients resumed treatment as per local standard of care. A safety follow up visit was done at Week 56.
Arm/Group | Mylan's Insulin Glargine | Lantus®
All-Cause Mortality (participants affected / at risk) | 2/280 | 1/278
Serious Adverse Events (participants affected / at risk) | 18/280 | 22/278
Other Adverse Events (participants affected / at risk) | 225/225 | 239/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mylan's Insulin Glargine (N=280) | Lantus® (N=278)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Malignant oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Generalized tonic-clonic seizure (Nervous system disorders) | 0 (0) | 2 (2)
Hypoglycaemic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Glomerulonephritis minimal lesion (Renal and urinary disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (7) | 10 (10)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mylan's Insulin Glargine (N=225) | Lantus® (N=239)
Hypertension (Vascular disorders) | 9 (9) | 6 (6)
Seasonal allergy (Immune system disorders) | 2 (4) | 3 (3)
Pyrexia (General disorders) | 5 (6) | 4 (4)
Oedema peripheral (General disorders) | 4 (4) | 3 (3)
Fatigue (General disorders) | 4 (4) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 4 (4)
Blood pressure increased (Investigations) | 0 (0) | 3 (3)
Tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 14 (20)
Carpal tunnel syndrome (Nervous system disorders) | 4 (5) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 0 (0)
Diabetic retinopathy (Eye disorders) | 2 (2) | 5 (5)
Nausea (Gastrointestinal disorders) | 10 (10) | 6 (8)
Diarrhoea (Gastrointestinal disorders) | 11 (12) | 4 (4)
Toothache (Gastrointestinal disorders) | 4 (7) | 5 (5)
Vomiting (Gastrointestinal disorders) | 6 (7) | 2 (3)
Microalbuminuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (13) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 154 (3045) | 170 (3184)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (6)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 25 (37) | 39 (58)
Upper respiratory tract infection (Infections and infestations) | 27 (38) | 33 (44)
Influenza (Infections and infestations) | 12 (12) | 12 (14)
Urinary tract infection (Infections and infestations) | 9 (13) | 10 (11)
Bronchitis (Infections and infestations) | 9 (9) | 8 (8)
Gastroenteritis (Infections and infestations) | 10 (10) | 6 (6)
Sinusitis (Infections and infestations) | 8 (10) | 8 (8)
Gastroenteritis viral (Infections and infestations) | 6 (6) | 7 (7)
Viral infection (Infections and infestations) | 5 (5) | 6 (6)
Pharyngitis (Infections and infestations) | 5 (5) | 2 (2)
Fungal infection (Infections and infestations) | 3 (3) | 3 (4)
Pharyngitis streptococcal (Infections and infestations) | 4 (6) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 5 (5)
Respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Onychomycosis (Infections and infestations) | 1 (1) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 3 (4)
Tonsilitis (Infections and infestations) | 3 (3) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days